CLINICAL TRIAL: NCT07357883
Title: Comparative Evaluation of Argan Oil as a Post-Operative Agent Versus Placebo Following Laser Gingival Depigmentation: A Randomized Controlled Clinical Trial
Brief Title: Effect of Topical Argan Oil on Healing After Laser Depigmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ghada Adayil (Other)
Responsible Party: Sponsor-Investigator, Ghada Adayil, Lecturer - Periodontology Department - Faculty of Dentistry - Cairo University., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 28-10-2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gingival Hyperpigmentation; Laser Depigmentation; Topical Argan Oil; Postoperative Gingival Healing
Keywords: Laser depigmentation; postoperative healing; topical argan oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Argan Oil (Experimental): Applied post-laser depigmentation
  Interventions: Procedure: Laser Depigmentation
- Reference placebo (Placebo Comparator): Identical placebo formulation
  Interventions: Procedure: Laser Depigmentation

INTERVENTIONS:
Procedure: Laser Depigmentation — Laser protocol:
  Diode laser, wavelength 810-980 nm, continuous mode, initiated fiber tip 400 µm, power 1.5-2 W.

SUMMARY:
Effect of Argan oil vs placebo on healing after laser depigmentation

DETAILED DESCRIPTION:
Evaluate the effect of Argan oil vs. placebo on post-operative healing after laser depigmentation. as well as Compare pain levels (VAS score), gingival pigmentation recurrence, and patient satisfaction between groups at predetermined follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 with moderate/severe physiological gingival pigmentation
* Good general and periodontal health.

Exclusion Criteria:

* Systemic diseases affecting healing (e.g., uncontrolled diabetes).
* Smokers or tobacco chewers.
* Pregnant/lactating women.
* Previous depigmentation procedures in the last 2 years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-10-29 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Effect of Argan oil | 14 days
  Evaluate the effect of Argan oil vs. placebo on post-operative Gingival healing

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 14 days
  Compare pain levels (VAS score) , gingival pigmentation recurrence, and patient satisfaction between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No